CLINICAL TRIAL: NCT05604534
Title: Assessing and Improving Quantitative Magnetic Resonance Imaging Metrics in Human Subjects
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000784; 000784-N
Record Dates: First submitted 2022-11-02; First posted 2022-11-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12-15

CONDITIONS: Normal Physiology
Keywords: MRI; Healthy Adult; Diffusion; DTI; Diffusion Tensor Imaging; Natural History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adult: Adults 18 years of age or older, in good general health

SUMMARY:
Background:

Magnetic resonance imaging (MRI), which uses strong magnets to get images of structures inside the body, is a valuable tool in modern medicine. But researchers are always looking for ways to improve this technology. To better understand how to use MRI to diagnose problems, researchers need to collect more data from scans of healthy people.

Objective:

To get MRI scans of healthy people to improve the measurements doctors can make from the images.

Eligibility:

People aged 18 years or older in good general health.

Design:

Participants will be screened. They will have a physical exam focused on their nervous system. They will complete questionnaires.

Participants will have at least 1 MRI scan. The target of the scan may be the brain, liver, prostate, breast, or other body part. Before the scan, participants will remove any metallic objects. They will lie on a narrow table that moves into a long, narrow tube. They may have special pads placed around them to help them remain still.

Participants will hear loud noises during the scan. They will get earplugs or earmuffs to wear to muffle the sound. They can communicate with the MRI technician and will have an emergency button to squeeze at any time if they want the scan to stop. The scan will take up to 2 hours.

Some participants may be asked to perform tasks on a computer screen during the scan.

Participants may return for up to 5 scans in 3 months. Some may have as many as 30 MRI visits per year. They may remain in the study for up to 2 years.

DETAILED DESCRIPTION:
Study Description:

Biomarkers are of fundamental importance for any clinical endeavor aimed at improving human health. The main objective of this protocol is to discover and investigate quantitative metrics obtained with non-invasive imaging techniques, primarily MRI, that could become potential biomarkers of the anatomical and physiological state of living human tissues, and to improve the experimental design of MRI acquisitions to enable reliable measurement of these quantitative metrics.

Objectives:

We will develop and optimize novel quantitative MRI (qMRI) techniques on normal, healthy volunteers, and investigate the accuracy and reproducibility of these novel techniques across time and across different MRI scanners.

Primary Objective: To improve the experimental design of MRI acquisitions to enable reliable measurement of quantitative metrics that are candidate biomarkers in human subjects.

Secondary Objectives: To assess the relative contributions of true inter-individual biological differences and experimental noise to the overall variability of the measured qMRI metrics.

Endpoints:

Primary Endpoint: Assessing the reproducibility of metrics derived from quantitative MRI data, evaluating the effects of acquisition modalities, such as experimental design, and choice of acquisition sequences and hardware, on the overall variability of these metrics.

Secondary Endpoints: Extracting the contributions of experimental design and biological variability to overall variability.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 years of age and older
* In good general health as evidenced by medical history
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Must have had a neurological physical exam as prescribed by NINDS policy. At the time of writing, this is required at least once every 2 years, and record of the exam should be in the medical record. This exam must be done prior to having MRI # 1. If deemed adequate by the Investigators, reports of examination by clinicians who are not Investigators on this study may be used. In addition, subjects must complete the most-recent version of the NMR safety screening form or NIH Radiology and IS MRI safety questionnaire when required at each visit.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Has any metal implant or objects of unknown identity or composition, or if it s known to be non-compatible with MRI, such as pacemakers, medication pumps, aneurysm clips, metallic prosthesis (such as heart valves or cochlear implants), certain orthopedic implants (pins and rods), shrapnel, or small metal fragments in the eye;
* Has claustrophobia to a degree that would preclude lying comfortably in the scanner for the duration of the examination;
* Cannot lie comfortably for up to 120 minutes;
* Has hearing problems which would make it difficult to tolerate scanner noise;
* Subjects with tattoos or permanent eye liner; liner; will not be excluded, however, tattoos carry a small risk of heating and burns. Therefore, each tattoo will be considered on a case by case basis, taking into account the age of the tattoo and the location of the tattoo on the subject s body.
* Has medical health problems such as pulmonary or airway disease, heart failure, coronary artery disease, which would require physiological monitoring during the scan;
* History of any medical condition that could result in an emergency medical situation while undergoing the MRI scan;
* For >7T: Has a ferromagnetic dental crown or a bridge.
* Non-English speakers are excluded as it is important that volunteers understand the complex instructions required to undergo an MRI procedure, and there is no direct benefit to participants.
* Pregnant women:

  * a) If a woman is pregnant at the time of enrollment, we will popstpone enrollment until she is no longer pregnant.
  * Participants will not remain on the study should they have a positive pregnancy test at a study visit.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18 years of age or older, in good general health, who live in the DMV area.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2041-03-31 (Estimated); Study Completion 2041-03-31 (Estimated)

PRIMARY OUTCOMES:
Assessing the reproducibility of metrics derived from quantitative MRI data, evaluating the effects of acquisition modalities, such as experimental design, and choice of acquisition sequences and hardware, on the overall variability of these met... | The completion of data collection
  For a given qMRI metric (e.g. mean diffusivity, T1, T2) under investigation and a given organ (e.g. brain, peripheral nerve, prostate) under investigation: 1) Map values of the metric under investigation throughout the organ 2) Measure the variability of the measured values in repeated scans on one MRI scanner 3) Measure the variability of the measured values acquired using proposed improvements in experimental design and document that a proposed improvement (e.g., improved pulse sequence acquisition, post processing technique) results in improved reproducibility.

SECONDARY OUTCOMES:
Extracting the contributions of experimental design and biological variability to overall variability. | The completion of data collection
  1) Extract the contributions of experimental noise to the overall variability through repeated scans in individual subjects 2) Using the experimental noise measurements from step 1, analyze differences across the study subject population to extract the true inter-individual biological differences.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo M Pierpaoli, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do plan to share IPD. we will share all IPD that results in a publication on a public repository, as required by most journals. the data will be de-identified and anonymized.

REFERENCES:
- [Background] Walker L, Curry M, Nayak A, Lange N, Pierpaoli C; Brain Development Cooperative Group. A framework for the analysis of phantom data in multicenter diffusion tensor imaging studies. Hum Brain Mapp. 2013 Oct;34(10):2439-54. doi: 10.1002/hbm.22081. Epub 2012 Mar 28. PMID 22461391
- [Background] Sadeghi N, Nayak A, Walker L, Okan Irfanoglu M, Albert PS, Pierpaoli C; Brain Development Cooperative Group. Analysis of the contribution of experimental bias, experimental noise, and inter-subject biological variability on the assessment of developmental trajectories in diffusion MRI studies of the brain. Neuroimage. 2015 Apr 1;109:480-92. doi: 10.1016/j.neuroimage.2014.12.084. Epub 2015 Jan 9. PMID 25583609
- [Background] Pierpaoli C. Quantitative brain MRI. Top Magn Reson Imaging. 2010 Apr;21(2):63. doi: 10.1097/RMR.0b013e31821e56f8. No abstract available. PMID 21613871
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000784-N.html